CLINICAL TRIAL: NCT02715583
Title: C-Acetate PET/CT Imaging to Evaluate Treatment Changes in Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 02816
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer Patients
MeSH Terms: interventions — carbon-11 acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with castrate resistant prostate cancer (CRPCA) with osseous metastatic disease. (Experimental): Patients with castrate resistant prostate cancer (CRPCA) with osseous metastatic disease planning to undergo Ra-223 therapy may be eligible for this study. Patients may participate in this study if they are at least 18 years of age, most participants will be receiving care at the clinical practices of the University of Pennsylvania.
  Positron emission tomography (PET/CT) imaging will use the investigational radiotracer [11C]acetate. Imaging will occur prior to Ra-223 therapy and after 2 cycles, in addition to standard of care 99mTcMDP bone scan at baseline and a research 99mTc-MDP bone scan post-therapy
  Patients will also undergo serial lab tests (PSA, and alkaline phosphatase levels). If these tests are done as part of clinical standard of care they will not need to be repeated for this study. Patients will be asked to complete a quality of life metric (short form of the McGill pain questionnaire) on the day of each PET/CT scan.
  Interventions: Drug: 11C-Acetate

INTERVENTIONS:
Drug: 11C-Acetate

SUMMARY:
Patients with castrate resistant prostate cancer (CRPCA) with osseous metastatic disease planning to undergo Ra-223 therapy may be eligible for this study. Positron emission tomography (PET/CT) imaging will use the investigational radiotracer [11C]acetate. Imaging will occur prior to Ra-223 therapy and after 2 cycles, in addition to standard of care 99mTcMDP bone scan at baseline and a research 99mTc-MDP bone scan post-therapy

DETAILED DESCRIPTION:
Our proposed study aims to use 11C-acetate PET/CT for evaluation of treatment response to Ra-223 dichrolide therapy. 11C-acetate has been shown to have superior detection of osseous and non-osseous metastatic lesions as compared to 18F-FDG PET/CT and 99Tc-MDP imaging. 11C-acetate is generally >80% sensitive for detection of metastatic lesions as compared to less than 70% for 18F-FDG PET/CT with higher tumor than tumor to background ratio14-19. The majority of interest in 11C-acetate PET/CT imaging is focused on the detection of distant metastatic disease in patients with biochemical relapse status post definitive local therapy18,20,21. In patients with 99Tc-MDP detected prostate bone metastases, Yu et al. have found that 11C-acetate PET/CT was superior to 18F-FDG PET/CT for evaluation of bone metastases treatment response regardless of hormonal or taxol based chemotherapy. In the Yu et al. pilot study, 11C-acetate PET/CT findings correlated with composite clinical designation of treatment response in 100% of patients22.

Our study will evaluate baseline standard uptake value (SUVmax) and change in SUVmax of 11C-acetate PET/CT at approximately 10 weeks weeks (+/- 3 weeks) , generally after two cycles of Ra-223 dichloride therapy. SUVmax will be recorded for a selected index lesion and an average of the 5 most 11C-acetate avid lesions, from the baseline scan. Evaluation of 11C-acetate uptake changes to therapy in this pilot study will allow sample size calculation for future trials correlating 11C-acetate changes to therapy to TTP, OS and symptomatic relief end points.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria at least 18 years of age
* History of biopsy proven or clinically documented castrate resistant prostate cancer which is metastatic to bone as assessed by medical record review.
* Patients selected for Ra-223 dichloride therapy for treatment of bone metastasis by their treating physician.
* Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* Not on current androgen deprivation therapy or plan for withdrawal of androgen deprivation therapy
* Cytotoxic chemotherapy within 4 weeks prior to study enrollment
* Systemic radioisotope therapy within 24 weeks prior to study enrollment
* Eminent or established cord compression as assessed by medical record review
* History of hemibody external radiotherapy as assessed by medical record review
* Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
* Serious or unstable medical or psychological comorbidities that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
* Documented visceral metastases or current lymphadenopathy > 3 cm by standard imaging (e.g. MRI, CT, ultrasound, FDG PET/CT)
* Only individuals (aged 18 or over) who can understand and give informed consent will be eligible to participate in this study. Individuals who are considered to be mentally disabled will not be recruited for this study. All subjects must be able to give informed consent. We will not be using specific methods to assess decisional capacity. Economically disadvantaged persons will not be vulnerable to undue influence, as this study offers no compensation. All individuals will be told that their choice regarding study participation will in no way change their access to clinical care. This should negate any undue influence or coercion. Women, children, fetuses, neonates, or prisoners are not included in this research study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03; Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Estimate the fold change in SUVmax () | 1 year
  • Estimate the fold change in SUVmax () of selected index lesions and the sum of SUVmax over the most 11C-acetate avid lesions, up to five, measured at pre and post Ra-223 dichrolide therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Pryma, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States